CLINICAL TRIAL: NCT00446641
Title: Phase 4 Study of Additional Cilostazol for Overcoming Biochemical Aspirin Resistance in the Chronic Stroke Patients
Brief Title: Overcome Biochemical Aspirin Resistance Through Cilostazol Combination
Acronym: ARCC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sun U. Kwon, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARCC
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Results first posted 2010-01-18 (Estimated); Last update posted 2010-01-18 (Estimated); Status verified 2009-11

CONDITIONS: Cerebral Infarction
Keywords: Infarction, Cerebral; Cilostazol; Aspirin Resistance
MeSH Terms: conditions — Cerebral Infarction | interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Cilostazol (Experimental): 100mg of Cilostazol twice a day
  Interventions: Drug: Cilostazol
- Placebo (Placebo Comparator): matching placebo to cilostazol
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Cilostazol — cilostazol 100mg twice a day for 4 weeks
  Other Names: pletaal
  Arms: 1 Cilostazol
Drug: placebo — placebo 1 tablet twice a day matching for cilostazol
  Other Names: matching placebo of cilostazol
  Arms: Placebo

SUMMARY:
This study will recruit 316 ischemic stroke patients taking aspirin.

They will be randomly assigned into cilostazol group or placebo group. Every patients will take 200mg of cilostazol a day or placebo for 1 month.

The primary outcome variable of this study is rate of biochemical aspirin resistance on the Ultra Rapid Platelet Function Assay-ASA.

DETAILED DESCRIPTION:
[Goal] To reveal the effect and safety of additional cilostazol for overcoming biochemical aspirin resistance.

[Trial Design] Double-Blind, Placebo-Controlled, Randomized, Multicenter Trial

[Participants] Ischemic stroke patients taking aspirin

[Methods]

* Double-Blind, Placebo-Controlled, Randomized, Multicenter Trial
* Investigational product: Cilostazol 200mg (100mg twice per day)
* Concomitant medication: Aspirin 100 mg per day
* Medication Duration: 1 month

[Outcome Variables]

Primary Outcome Variable:

• the proportion of patients with aspirin reaction units (ARUs) values ≥550 on the Ultra Rapid Platelet Function Assay-ASA

Secondary outcome variables:

* the proportion of patients with ARUs values ≥500 on the Ultra Rapid Platelet Function Assay-ASA
* ARUs values
* Bleeding time (BT)
* Fatal or major bleeding complications
* Any bleeding complications

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic cerebral infarction documented on MRI or CT
* More than 35 years of age
* Patients taking aspirin 100mg a day for 2 weeks or more before randomization

Exclusion Criteria:

* Patients taking any antiplatelets other than aspirin within 2 weeks before randomization
* Patients taking any anticoagulants within 2 weeks before randomization
* Patients taking thrombolytic therapy within 2 weeks before randomization
* Patients taking any NSAIDs within 2 weeks before randomization
* Patients who need to take NSAIDs regularly (e.g. rheumatic arthritis).
* Bleeding diathesis
* Chronic liver disease (ALT > 100 or AST > 100) or chronic renal disease (creatinine > 3.0mg/dl)
* Anemia (hemoglobin < 10mg/dl) or thrombocytopenia (platelet count less than 100,000/mm3)
* Pregnant or lactating patients
* Patients scheduled for angioplasty or revascularization procedures within 4 weeks
* Patients scheduled for any surgery or invasive procedures within 4 weeks
* Patients having acute coronary syndrome

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2007-03; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sun U Kwon, MD. PhD., Principal Investigator — Asan Medical Center, Univsersity of Ulsan, Medical College
Locations (4):
- South Korea (4):
  - Jae-Kwan Cha, Busan, Busan
  - Eulji University Hospital, Daejeon
  - Kangdong Sacred Heart Hospital, Hallym University, Seoul
  - Asan Medical Center, Seoul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 244 patients with subacute or chronic ischemic stroke were recruited from outpatient clinics of 5 comprehensive stroke centers of Korea
Pre-assignment Details: Patients with aspirin therapy were recruited due to subacute or chronic ischemic stroke.
  The patients should have taken aspirin 100mg per day at least 2 weeks before randomization
Groups:
- Cilostazol: Cilostazol 100mg twice per day
Period: Overall Study
Arm/Group | Cilostazol | Placebo
Started | 125 | 119
Completed | 108 | 109
Not Completed | 17 | 10
Not completed — Withdrawal by Subject | 8 | 3
Not completed — poor compliance | 8 | 6
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cilostazol | Placebo | Total
Number analyzed (Participants) | 125 | 119 | 244
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 71 | 146
  >=65 years | 50 | 48 | 98
Age Continuous [Mean (Standard Deviation); unit: years] | 61.24 (10.198) | 62.83 (9.963) | 62.02 (10.095)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 41 | 77
  Male | 89 | 78 | 167
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 125 | 119 | 244

OUTCOME MEASURES:

1. Primary Outcome: Aspirin Resistance (ARU ≥ 550)
Description: The number of patients with aspirin reaction units (ARUs) values ≥ 550 on the Ultra Rapid Platelet Function Assay-ASA among the recruited patients
Time Frame: 4 weeks after treatment
Measure: Number; unit: participants
Arm/Group | Cilostazol | Placebo
Number analyzed (Participants) | 108 | 109
participants | 9 | 11
Statistical Analysis 1: Comparison: Cilostazol vs Placebo; We assumed that the prevalence of AR would be 12 % among ischemic stroke patients who were treated with aspirin 100 per day. The prevalence could be reduced to 4% with additional cilostazol therapy; Test type: Superiority or Other; p = 0.654, Chi-squared; Odds Ratio (OR) = 0.82

2. Secondary Outcome: Aspirin Resistance (ARU ≥ 500)
Description: The number of participants with ARUs values ≥500 on the Ultra Rapid Platelet Function Assay-ASA; ARUs values
Time Frame: 4 weeks after reatment
Measure: Number; unit: participants
Arm/Group | Cilostazol | Placebo
Number analyzed (Participants) | 108 | 109
participants | 20 | 28

3. Secondary Outcome: Bleeding Time (BT)
Description: for evaluation of the extent of the bleeding time prolongation by additional cilostazol
Time Frame: 4 weeks after reatment
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Cilostazol | Placebo
Number analyzed (Participants) | 108 | 109
seconds | 113 (38.5) | 106 (34.2)

4. Secondary Outcome: Fatal or Major Bleeding Complications;
Description: Fatal or life-threatening bleeding was defined as any fatal bleeding event, a drop in hemoglobin of ≥ 50g/L, or significant hypotension with need for inotropic agents, symptomatic intracranial hemorrhage, or transfusion of ≥ 4 units of red-blood cells or equivalent amount of whole blood. Major bleeding was defined as significantly disabling bleedings, intraocular bleeding leading to significant visual loss, or bleeding requiring transfusion of ≤ 3 units of red-blood cells or equivalent amount of whole blood
Time Frame: events ocurred during study medication after randomization
Measure: Number; unit: participants
Arm/Group | Cilostazol | Placebo
Number analyzed (Participants) | 108 | 109
participants | 0 | 0

5. Secondary Outcome: Any Bleeding Complications
Description: any bleeding events causing medical attention
Time Frame: events ocurred during study medication after randomization
Measure: Number; unit: participants
Arm/Group | Cilostazol | Placebo
Number analyzed (Participants) | 108 | 109
participants | 0 | 0

6. Secondary Outcome: Difference of Post-treatment ARU and Baseline ARU
Description: summation of change of ARU (posttreatment ARU - baseline ARU) of individual patients
Time Frame: baseline ARU measured at the randomization and post-treatment ARU measured at the 4weeks treatment with study medication
Measure: Mean (Standard Deviation); unit: change of ARU measured
Arm/Group | Cilostazol | Placebo
Number analyzed (Participants) | 108 | 109
change of ARU measured | -7.8 (77.6) | 12.1 (71.1)

7. Secondary Outcome: Post-treatment ARU
Description: mean of ARU value of individual participants after 4 weeks treatment
Time Frame: after 4 weeks treatment
Measure: Mean (Standard Deviation); unit: ARU
Arm/Group | Cilostazol | Placebo
Number analyzed (Participants) | 108 | 109
ARU | 454.8 (52.8) | 473.6 (63.9)

ADVERSE EVENTS:
Arm/Group | Cilostazol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/125 | 0/119
Other Adverse Events (participants affected / at risk) | 7/125 | 2/119
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cilostazol (N=125) | Placebo (N=119)
headache (Nervous system disorders) | 7 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No